CLINICAL TRIAL: NCT04217590
Title: A Phase 3b, Multicentre, Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Reduce Incidence of Pre-Dialysis Hyperkalaemia With Sodium Zirconium Cyclosilicate in Chinese Subjects
Brief Title: Reduce Incidence of Pre-Dialysis Hyperkalaemia With Sodium Zirconium Cyclosilicate in Chinese Subjects
Acronym: DIALIZE China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9485C00001
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; Streptozocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium Zirconium Cyclosilicate (SZC) (Experimental): Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of SZC 5g depending on dose level assigned to a patient per non-dialysis days.
  Interventions: Drug: Sodium Zirconium Cyclosilicate
- Placebo (Placebo Comparator): Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of Placebo depending on dose level assigned to a patient per non-dialysis days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of SZC 5g depending on dose level assigned to a patient per non-dialysis days.
  Other Names: SZC; Lokelma; ZS
  Arms: Sodium Zirconium Cyclosilicate (SZC)
Drug: Placebo — Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of Placebo depending on dose level assigned to a patient per non-dialysis days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sodium Zirconium Cyclosilicate (SZC), as well as the appropriateness of the dosing mechanism, in Chinese end-stage renal disease (ESRD) patients on chronic haemodialysis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to determine the safety and efficacy of SZC in ESRD subjects with hyperkalaemia and on stable haemodialysis. This study consists of a screening period, an 8-week randomized treatment period, and a follow-up period. Approximately 134 stable haemodialysis subjects with persistent pre-dialysis hyperkalaemia will be enrolled in the study across research sites in China.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
2. Subject must be ≥ 18 years of age inclusive, at the time of signing the informed consent form.
3. Subjects must have haemodialysis access consisting of an arteriovenous fistula, AV graft, or tunnelled (permanent) catheter which is expected to remain in place for the entire duration of the study.
4. Receiving haemodialysis (or hemodiafiltration) 3 times a week for treatment of end-stage renal disease (ESRD) for at least 3 months before randomization.
5. Pre-dialysis S-K > 5.4 mmol/L after long inter-dialytic interval and > 5.0 mmol/L after at least one short inter-dialytic interval during screening (as assessed by central lab).
6. Prescribed dialysate K concentration ≤ 3 mmol/L during screening.
7. Sustained Qb ≥ 200 ml/min and spKt/V ≥ 1.2 (or URR ≥ 63) on stable haemodialysis / haemodiafltration prescription during screening with prescription (time, dialyzer, blood flow [Qb], dialysate flow rate [Qd] and bicarbonate concentration) expected to remain unchanged during study.
8. Subjects must be receiving dietary counselling appropriate for ESRD subjects treated with haemodialysis / haemodiafiltration as per local guidelines, which includes dietary potassium restriction.

Exclusion Criteria:

1. Myocardial infarction, acute coronary syndrome, stroke, seizure or a thrombotic / thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism, but excluding vascular access thrombosis) within 12 weeks prior to randomization.
2. Pseudohyperkalaemia secondary to haemolyzed blood specimen (this situation is not considered screening failure, sampling or full screening can be postponed to a later time as applicable).
3. Diagnosis of rhabdomyolysis during the 4 weeks preceding randomization.
4. Presence of cardiac arrhythmias or conduction defects that require immediate treatment.
5. Any medical condition, including active, clinically significant infection or liver disease, that in the opinion of the investigator or Sponsor may pose a safety risk to a subject in this study, which may confound safety or efficacy assessment and jeopardize the quality of the data, or may interfere with study participation.
6. History of QT prolongation associated with other medications that required discontinuation of that medication; congenital long QT syndrome or QTc(f) > 550 msec; uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication or with transient atrial fibrillation associated with dialysis or peridialytic period are permitted.
7. Subjects treated with sodium polystyrene sulfonate (e.g. SPS, Kayexalate, Resonium), calcium polystyrene sulfonate (CPS, Resonium calcium) or patiromer (Veltassa) within 7 days before screening or anticipated in requiring any of these agents during the study.
8. Participation in another clinical study with an investigational product administered in the last 1 month before screening.
9. Haemoglobin < 9 g/dL on screening (as assessed on Visit 1).
10. Laboratory diagnosis of hypokalaemia (K < 3.5 mmol/L), hypocalcemia (Ca < 8.2 mg/d or albumin-corrected Ca < 8.0 mg/dL if the latter is used in local practice), hypomagnesemia (Mg < 1.7 mg/dL) or severe acidosis (serum bicarbonate 16 mEq/L or less) in the 4 weeks preceding randomization.
11. Severe leukocytosis (> 20 × 109/L) or thrombocytosis (≥ 450 × 109/L) during screening.
12. Polycythaemia (Hb > 14 g/dL) during screening.
13. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
14. Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.
15. Previous randomisation in the present study.
16. For women only - currently pregnant (confirmed with positive pregnancy test or uterine ultrasound if pregnancy test is questionable) or breast-feeding.
17. Females of childbearing potential, unless using contraception as detailed in the protocol or sexual abstinence.
18. Lack of compliance with haemodialysis prescription (both number and duration of treatments) during the two-week period preceding screening (100% compliance required).
19. Subjects unable to take investigational product drug mix.
20. Scheduled date for living donor kidney transplant.
21. Subjects with a life expectancy of less than 6 months.
22. Known hypersensitivity or previous anaphylaxis to SZC or to components thereof.
23. History of alcohol or drug abuse within 2 years prior to randomization.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Ni, Principal Investigator — Department of Nephrology, Renji Hospital, School of Medicine, Shanghai Jiaotong University, China.
Locations (19):
- China (19):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Dongguan
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ni Z, Lu R, Xu X, Bian X, Zhou Z, Yang J, Luo Q, Chen M, Chen C, Sun X, Yu L, He Q, Jiang H, Yuan W, Li Y, Zhou R, Wang J, Zhang X, Zuo L, Meng X, Chang Z, Zhao J, Wessman P, Xiang P; DIALIZE China Study Group. DIALIZE China: A Phase IIIb, Randomized, Placebo-Controlled Study to Reduce Predialysis Hyperkalemia With Sodium Zirconium Cyclosilicate in Chinese Patients. Clin Ther. 2023 Jul;45(7):633-642. doi: 10.1016/j.clinthera.2023.04.014. Epub 2023 Jun 27. PMID 37385905
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9485C00001&attachmentIdentifier=1c10b684-b39c-4155-a455-25f3ec2a77c2&fileName=CSP_Redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9485C00001&attachmentIdentifier=5e2a8f35-b41e-4685-899a-6ffa81781403&fileName=Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9485C00001&attachmentIdentifier=8fff0273-c810-405f-9ee1-2145eff8f169&fileName=CSR_synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been completed and was conducted in 37 centres across China. 281 subjects were screened and 134 randomised subjects (67 per treatment group).
Pre-assignment Details: Eligbile Chinese subjects with end-stage renal disease (ESRD) on stable haemodialysis were randomly assigned to either sodium zirconium cyclosilicate (SZC) or placebo in a 1:1 ratio.
Groups:
- Sodium Zirconium Cyclosilicate (SZC); Placebo: Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose).
  Single dose contains 1 to 3 sachets that should be suspended in 45 mL of water by patient and administered on non-dialysis days.
Period: Overall Study
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Started | 67 | 67
Completed | 63 | 64
Not Completed | 4 | 3
Not completed — Other | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on all patients in the full analysis set (FAS), which comprised all patients randomized. Patients were included in the analysis in the treatment arm to which they were randomized, regardless of the treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (11.32) | 54.5 (11.36) | 54.7 (11.30)
Age, Customized [Count of Participants; unit: Participants]
  Age group (years): <50 years | 20 | 22 | 42
  Age group (years): >=50 - <65 years | 33 | 33 | 66
  Age group (years): >=65 -<85 years | 14 | 11 | 25
  Age group (years): >=85 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 67 | 67 | 134

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: A subject was considered to be a responder if, during the evaluation period, they maintained a pre-dialysis serum potassium (S-K) between 4.0 and 5.0 mmol/L on at least 3 out of 4 dialysis treatments following the long inter-dialytic interval (LIDI) and did not receive rescue therapy. Subjects with no data during the evaluation period were classified as non-responders. The S-K levels used for this analysis were based on the measurements obtained by the central laboratory.
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 67 | 67
Participants | 25 | 7
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 5.10, 95% CI 2-sided [1.90 to 15.12] — The CI for OR is calculated as an exact CI. An OR > 1 favours SZC

2. Secondary Outcome: Maximum Pre-dialysis S-K Values After SIDI and LIDI Below or Equal to 5.5 mmol/L During Evaluation Period
Description: Probability of maintaining maximum S-K value <= 5.5 mmol/L was evaluated. Each subject's maximum pre-dialysis S-K at long inter-dialytic interval (LIDI) and short inter-dialytic interval (SIDI) visits during the evaluation period were categorised into <= 5.5 or > 5.5 mmol/L. Missing S-K values including those omitted due to coinciding with rescue therapy use or records omitted that are not true LIDI (i.e. records which do not occur >= 55 hours after the previous dialysis starting time) were imputed using multiple imputation (MI).
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Number; unit: Probability
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 67 | 67
Probability | 0.54 | 0.15
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; The OR, 95% CI and p-value are obtained from a pooled logistic regression model after multiple imputation (MI) of missing pre-dialysis S-K values; Odds Ratio (OR) = 6.41, 95% CI 2-sided [2.64 to 15.55] — An OR > 1 favours SZC

3. Secondary Outcome: Pre-dialysis S-K After LIDI Between 3.5 and 5.5 mmol/L During the Evaluation Period
Description: Probability of all S-K values between 3.5 and 5.5 mmol/L was evaluated. Subjects were categorised to either having all pre-dialysis LIDI values between 3.5 and 5.5 mmol/L during the evaluation period or not. Missing S-K values including those omitted due to coinciding with rescue therapy use or records omitted that are not true LIDI (i.e. records which do not occur >= 55 hours after the previous dialysis starting time) were imputed using multiple imputation (MI).
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Number; unit: Probability
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 67 | 67
Probability | 0.58 | 0.17
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 6.41, 95% CI 2-sided [2.71 to 15.12] — An OR > 1 favours SZC

4. Secondary Outcome: Instances of Pre-dialysis S-K After LIDI Between 4.0 and 5.0 mmol/L During the Evaluation Period
Description: The probability of maintaining instances of pre-dialysis S-K between 4.0 and 5.0 mmol/L (normokalaemia) was evaluated at each LIDI visit during the evaluation period, by categorisation of pre-dialysis S-K into values between 4.0 and 5.0 mmol/L or not. Values coinciding with rescue therapy or not true LIDI (i.e. records which do not occur >= 55 hours after the previous dialysis starting time) were excluded.
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Number; unit: Probability
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 63 | 64
Probability | 0.48 | 0.17
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Generalised linear mixed model (GLMM); The p-value was obtained from a test of equality of odds ratios; Odds Ratio (OR) = 4.41, 95% CI 2-sided [2.53 to 7.67] — The OR was obtained from GLMM model with random intercept and logit link. Treatment, visit, visit by treatment interaction and baseline were specified as fixed effects. An OR > 1 favours SZC

5. Secondary Outcome: Expected Number of Normokalaemic (S-K 4.0-5.0 mmol/L) Instances
Description: The expected number of normokalemic instances is the sum of the probabilities of normokalaemic instance at each visit during the evaluation period. Normokalaemic is defined as S-K between 4.0 and 5.0 mmol/L.
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Number; unit: Sum of probabilities
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 63 | 64
Sum of probabilities | 1.91 | 0.70
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [0.77 to 1.64] — Endpoint analysed with Generalised linear mixed model. The CI for the mean difference was calculated by bootstrapping. A mean difference > 0 favours SZC

6. Secondary Outcome: Instances of Potassium Gradient of < 3.0 mmol/L After LIDI During the Evaluation Period
Description: The probability of maintaining instances of potassium gradient of < 3.0 mmol/L was evaluated at each LIDI visit during the evaluation period, by categorisation of potassium gradient into < 3.0 or >=3.0 mmol/L. Values coinciding with rescue therapy or not true LIDI (i.e. records which do not occur >= 55 hours after the previous dialysis starting time) were excluded.
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks.
Population: Full analysis set
Measure: Number; unit: Probability
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 63 | 64
Probability | 0.52 | 0.16
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Generalised linear mixed model (GLMM); The p-value was obtained from a test of equality of odds ratios; Odds Ratio (OR) = 5.82, 95% CI 2-sided [3.15 to 10.73] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Includes adverse events that occurred from time of randomization throughout the treatment period and follow-up period, up to end of study visit (Day 71 +/- 3 days) or premature study discontinuation visit.
Description: Safety Analysis Set (All randomized subjects who received at least 1 dose of investigational product, SZC or placebo. N=66 for SZC, N=67 for Placebo). Subjects excluded from the Safety Analysis Set (n=1 for SZC, n=0 Placebo) did not receive treatment.
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/67
Serious Adverse Events (participants affected / at risk) | 6/66 | 8/67
Other Adverse Events (participants affected / at risk) | 24/66 | 25/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) (N=66) | Placebo (N=67)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhagic gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) (N=66) | Placebo (N=67)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (10) | 6 (7)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Dialysis hypotension (Vascular disorders) | 3 (17) | 4 (10)
Hypotension (Vascular disorders) | 3 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (8) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT04217590/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT04217590/SAP_001.pdf